CLINICAL TRIAL: NCT05625425
Title: Virtual Reality Interventions to Stimulate Capabilities for Learning and Retrieval of High-Fidelity Memory
Brief Title: Wayfinding Intervention and Long-Term Memory
Acronym: Quest-Tablet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-27586-B
Record Dates: First submitted 2022-11-10; First posted 2022-11-23 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Long-Term Memory Decline; Mild Cognitive Impairment
Keywords: amnestic MCI without dementia; cognitive training; cognitive aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: After recruitment, participants are randomly assigned to treatment arms. Participants and experimenters with whom participants interact during the experiments are blind to the purpose of the randomly-assigned arm. First-level analysis performed blind to participant's treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LabyrinthVR Scoot (Experimental): Multi-session cognitive intervention with VIVE high-resolution head-mounted display virtual reality computer game that presents an adaptive spatial wayfinding challenge. Game movement via handheld controllers.
  Interventions: Behavioral: LabyrinthVR software
- Placebo Controls (Placebo Comparator): Multi-session cognitive intervention with handheld tablet or wireless virtual reality headset presentation of commercially available, narrative computer games.
  Interventions: Behavioral: Placebo Games software
- Labyrinth Tablet (Experimental): Multi-session cognitive intervention with tablet computer, displaying 2.5D version of Labyrinth game in an adaptive spatial wayfinding challenge. Game movement via on-screen control buttons.
  Interventions: Behavioral: Labyrinth Tablet software
- Labyrinth VR wireless (Experimental): Multi-session cognitive intervention with QUEST head-mounted display virtual reality computer game using wireless technology to present an adaptive spatial wayfinding challenge. Game movement via handheld controllers.
  Interventions: Behavioral: Labyrinth VR wireless

INTERVENTIONS:
Behavioral: LabyrinthVR software — Head-mounted display virtual reality game designed to induce environmental enrichment in an adaptive, highly engaging regimen of wayfinding in novel urban and village neighborhoods.
  Arms: LabyrinthVR Scoot
Behavioral: Placebo Games software — Commercially-available, narrative computer games marketed as cognitively enriching. Can be tablet-based or wireless VR headset-based.
  Arms: Placebo Controls
Behavioral: Labyrinth Tablet software — Tablet computer playing Labyrinth spatial wayfinding game in 2.5D
  Arms: Labyrinth Tablet
Behavioral: Labyrinth VR wireless — Wireless head-mounted display virtual reality game designed to induce environmental enrichment in an adaptive, engaging regimen of wayfinding in novel urban and village neighborhoods.
  Arms: Labyrinth VR wireless

SUMMARY:
Therapeutic treatment is yet available for declining memory, which is an impairment affecting the quality of life for many older adults and patients with cognitive impairment. Cognitive training with an immersive video game promises to drive hippocampal-cortical plasticity and associated gains that can restore memory capability or provide therapeutic treatment for memory deficits.

DETAILED DESCRIPTION:
A hallmark of higher cognition is the capability for flexible association of diverse bits of information stored in memory, such that experiences can be remembered in detailed and distinct terms (i.e., high-fidelity long-term memory). Interventions capable of sustaining improved learning and flexible association of new information into long-term memory (LTM) have shown promising pilot results, and further development is expected to find treatments to attenuate the decline of high-fidelity LTM in normal aging or provide therapeutic treatment for patients with cognitive impairment without dementia (i.e., MCI).

This project applies a translational neuroscience approach in further development of a cognitive training intervention that targets sustained improvement in capabilities for long-term memory (LTM) and cognitive control. Treatments use commercially available head-mounted display Virtual Reality (VR) technology and tablet computers to present a deeply immersive spatial wayfinding video game.

Based on preliminary results, the hypothesis is that immersion in a game to navigate errands through unfamiliar, visually complex neighborhoods (i.e., wayfinding) will be an effective means to environmental enrichment, which refers to a process whereby new and complex experiences bring change to brain and behavior. Research in humans shows that learning a new, enriched environment spurs the healthy function of the hippocampus and supports lifelong neurogenesis. Adult-borne hippocampal neurogenesis has been linked as the neurobiological basis for the formation of new, high-fidelity memories.

The significance of this project includes functionality for remote training procedures (i.e., at home). The availability for participants to complete some of the experiment procedures at home will expand enrollment opportunities and prove the practicality of the intervention outside of a clinical setting.

The Labyrinth spatial wayfinding game uses 3D and 2.5D computer graphics tools to present dozens of levels of adaptive challenge and deliver a dynamic, engaging experience for participants throughout the training regimen. In this project, participants will effect game movement using hand controllers while playing the game in a seated position.

For each participant, pre- and post-training assessments will occur promptly before and after their 15 to 20-hour training regimen. Cognitive outcome measures will assess capabilities for high-fidelity LTM retrieval and control of sustained visual attention, and some measures will include collection of associated functional MRI (fMRI) and structural MRI data.

Effectiveness of the wayfinding game intervention will be evidenced by post-training improvements in retrieval of high-fidelity LTM and cognitive control capabilities. FMRI results associated with the measured cognitive improvements will localize changes in functional brain networks that support gains in memory capabilities. Structural MRI measures will assess morphometric and volumetric changes from pre- to post-training assessments.

ELIGIBILITY:
Inclusion Criteria:

* fluent speakers of English
* completed 12 or more years of education
* normal or corrected-to-normal vision
* dexterity to comfortably operate the scanner-compatible response box
* freedom from physical and neurological conditions contra-indicated for fMRI
* must confirm physical stamina and comfort for semi-weekly brisk 30-minute walks on level ground

Exclusion Criteria:

* use of psychotropic medications
* history of concussions or dizziness, vestibular or balance problems
* significant discomfort with virtual reality experiences

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
MDT change in mnemonic discrimination | baseline immediately before (T1) and post-assessment immediately after training regimen is completed (T2) providing for a composite score T2-T1
  Training-related change in Mnemonic Discrimination Task (MDT) score. MDT tests recognition memory for pairs of common objects (i.e., targets and lures), measuring the variable of the number of images identified as old (studied) or new (novel), and reports a composite index score (0.00 to 1.00) for accuracy post-training (T2) versus baseline (T1)
TOUR change in recall | baseline immediately before (T1) and post-assessment immediately after training regimen is completed (T2) providing for a composite score T2-T1
  Training-related change in recall of number of details in autobiographical memory from a narrated urban tour, such that a composite parametric score shows how many specific details were recalled post-training (T2) versus baseline (T1)
Volumetric-based brain morphometry for gray and white matter | collected in association with Outcome 1, at baseline immediately before (T1) and post-assessment immediately after training regimen is completed (T2)
  Structural MRI T1 data will be analyzed in terms of volumetric-based morphometry, measuring the variables of cortical area.
Task-based cortical functional connectivity associated with mnemonic discrimination capability and in control of sustained visual attention | collected in association with Outcome 1, at baseline immediately before (T1) and post-assessment immediately after training regimen is completed (T2)
  functional MRI data will be analyzed in terms of beta-series correlations between co-active cortical regions of interest, measuring the variable of correlation of inter-trial variability across brain regions

SECONDARY OUTCOMES:
Remote Cognitive Module (RCM) | baseline immediately before training regimen begins
  A tablet application using a speech-text interface to administer neuropsychological tests comparable to CVLT-II verbal memory, verbal fluency, digit span and Trail Making Test-B. Measured variables are target words remembered

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Wais, PhD, Principal Investigator — Neuroscape, Department of Neurology
Locations (1):
- UCSF Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No